CLINICAL TRIAL: NCT04599647
Title: Expanded Access Protocol for the Treatment of Glioblastoma With PVSRIPO
Brief Title: EAP for the Treatment of Glioblastoma With PVSRIPO
Status: No longer available | Type: Expanded Access
Sponsor: Istari Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PVSRIPO GBM EAP
Record Dates: First submitted 2020-10-16; First posted 2020-10-23 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: PVSRIPO — PVSRIPO (5x10^7 TCID50) delivered intratumorally via convection enhanced delivery (CED).

SUMMARY:
This is an open-label, single-arm, non-randomized, intermediate-sized expanded access study evaluating the safety, efficacy, and tolerability of PVSRIPO delivered via intratumoral infusion, in subjects with glioblastoma (GBM) who are ineligible to participate in clinical study with PVSRIPO that is currently open to enrollment.

ELIGIBILITY:
As a general principle, subjects eligible for access must:

* Have a serious or life-threatening condition;
* Have no appropriate, comparable, or satisfactory alternative treatment available, or such alternatives have been tried without clinical success, including clinical studies; and
* Be unable to participate in a PVSRIPO clinical trial that is currently open to enrollment.

Subjects are eligible if all of the following criteria are met:

1. Age ≥ 18 years at time of consent.
2. The subject is able and willing to provide written informed consent.
3. Subjects with:

   1. Prior histologically confirmed supratentorial GBM based on imaging studies with measurable disease (≥ 1 cm of contrast-enhancing tumor; multifocal acceptable if total enhancing disease burden considered acceptable); OR
   2. Subjects with GBM > 5.5 cm in diameter (these are excluded from current clinical studies of PVSRIPO), but for whom PVSRIPO is judged by Investigator to be appropriate for treatment. Such cases may include subjects with large resection cavities with residual infusible tumor, where the cavity allows space for expansion of peritumoral edema (PTE); OR
   3. Subjects with recurrent GBM (rGBM) who benefitted from prior PVSRIPO treatment; OR
   4. Subjects with GBM who do not meet eligibility for a clinical trial of PVSRIPO currently open to enrollment, but who would otherwise benefit from treatment. If appropriate, comparable or satisfactory alternative treatments approved for GBM must have been tried without clinical success, or in the opinion of the Investigator the subject is not a good candidate for those treatments but is anticipated to potentially benefit from PVSRIPO treatment without additional risk.
4. Before catheter placement based on screening MRI and at the time of catheter placement via CT prior to infusion, neurosurgical investigator should confirm placement of infusion catheter within or through the progressive enhancing tumor is feasible and at a safe distance relative to eloquent brain function, with the tip of the catheter being placed within these guidelines:

   1. Within the enhancing portion or in the vicinity of enhancement of target lesion (ie, infiltrative disease)
   2. ≥ 0.5 cm from ventricles
   3. ≥ 1 cm deep into the brain
   4. ≥ 0.5 cm from the corpus callosum

   Any changes from the above catheter tip placement guidelines require discussion and prior approval from the Sponsor.
5. Women of childbearing potential must have a negative urine or serum (Beta-Human Chorionic Gonadotropin, β-hCG) pregnancy test prior to PVSRIPO infusion.
6. Women and men in the study, and female partners of men in the study, must use highly effective birth control for 6 months after the last dose of PVSRIPO.
7. Karnofsky Performance Status (KPS) Score ≥ 70%.
8. Undergone prior vaccination against PV and received a boost immunization with trivalent IPOL® (Sanofi-Pasteur SA) at least 1 week, but less than 6 weeks, prior to administration of PVSRIPO (within 6 months of PVSRIPO retreatment). Note: Patients who are unsure of their prior vaccination status/who have not been vaccinated must provide proof of vaccination and/or evidence of anti-PV immunity prior to enrollment, as applicable.
9. Prior to biopsy (if required)/catheter placement, the following must be met: Platelet count ≥ 100,000/µL unsupported is necessary for eligibility; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/µL is required for the subject to undergo biopsy/catheter insertion, which can be attained via platelet transfusion (ie, supported).

Subjects with any of the following are excluded:

1. Women who are pregnant or breast-feeding.
2. Have an impending, life-threatening cerebral herniation syndrome, based on the assessment of the institution's neurosurgeons, and/or designee(s).
3. Have severe, active co-morbidity, defined as follows:

   1. Have an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C).
   2. Have known immunosuppressive disease or known human immunodeficiency virus infection.
   3. Have unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4).
   4. Have known lung (forced expiratory volume in the first second of expiration [FEV1] < 50%) disease or uncontrolled diabetes mellitus.
   5. Have an albumin allergy or serious gadolinium allergy/anaphylaxis.
4. Local laboratory values within two weeks of biopsy/catheter placement that meet any of the following:

   1. Prothrombin (PT) and activated Partial Thromboplastin Times (aPTT) > 1.5 × upper limit of normal (ULN)
   2. Total bilirubin, serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), alkaline phosphatase > 2.5 × ULN
   3. Neutrophil count < 1000/µL
   4. Hemoglobin < 9.0 g/dL
   5. Creatinine > 1.2 x ULN
5. Previous history of neurological complications due to PV infection.
6. Not recovered from the toxic effects of prior chemo- and/or radiation therapy, if applicable. Guidelines for this recovery period are dependent upon the specific therapeutic agent received; the following are excluded relative to planned PVSRIPO treatment:

   1. Tumor treating fields: ≤ 1 week
   2. Chemotherapy or bevacizumab: ≤ 4 weeks (except for nitrosourea and lomustine: ≤ 6 weeks)
   3. Metronomic dosed chemotherapy, such as daily temozolomide, etoposide or cyclophosphamide: ≤ 1 week
7. Prior, unrelated malignancy deemed unstable by the Investigator, except for cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin.
8. May not have received immunotherapy ≤ 4 weeks prior to PVSRIPO treatment unless the subject has recovered from side effects of such therapy, as determined by the Investigator.
9. May not be less than 12 weeks from radiation therapy of the brain unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation.
10. Evidence of diffuse subependymal or leptomeningeal disease or tumor in the brainstem, cerebellum, or spinal cord.
11. Undetectable anti-tetanus toxoid immunoglobulin G (IgG) (except for retreatment). If undetectable, a tetanus booster will be required at least 1 week, but less than 6 weeks, prior to administration of PVSRIPO.
12. Known history of agammaglobulinemia.
13. On ≥ 4 mg/day of dexamethasone within the 2 weeks prior to admission for PVSRIPO infusion.
14. Worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups).
15. Concomitant disease, condition, or disorder that deems the subject unsuitable for treatment with PVSRIPO in the opinion of the Investigator.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States